CLINICAL TRIAL: NCT07301294
Title: Microbiological Characteristics of Biofilm on Double J Ureteral Stents After Lithotripsy: A Randomized Controlled Trial
Brief Title: Microbiological Characteristics of Biofilm on Double J Ureteral Stents After Lithotripsy.
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Menoufia University (Other)
Responsible Party: Principal Investigator, Ammar Fathi Mohamed AlOrabi, Dr, Menoufia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Biofilm of DJ stent
Record Dates: First submitted 2025-12-22; First posted 2025-12-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Double J Stent
Keywords: DJ stent; Double J stent; ureteric stent; Biofilm; Mucolytic; Linezolid
MeSH Terms: interventions — Linezolid; Acetylcysteine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Control group (No Intervention): Patients of this group will receive no medications
- Antibiotic group (Active Comparator): Patients of this group will receive Linezolid.
  Interventions: Drug: Linezolid (LZD)
- Mucolytic group (Active Comparator): Patients of this group will receive N-Acetylcysteine.
  Interventions: Drug: N-Acetyl Cysteine (NAC)
- Combination group (Active Comparator): Patients of this group will receive both Linezolid and N-Acetylcysteine.
  Interventions: Drug: Linezolid (LZD); Drug: N-Acetyl Cysteine (NAC)

INTERVENTIONS:
Drug: Linezolid (LZD) — Linezolid 600 mg, oral, twice daily, for 7 days.
  Arms: Antibiotic group; Combination group
Drug: N-Acetyl Cysteine (NAC) — N-Acetyl cysteine 600 mg, oral, once daily, for 30 days.
  Arms: Combination group; Mucolytic group

SUMMARY:
Indwelling Double J (DJ) ureteral stents are commonly used following lithotripsy to ensure adequate urinary drainage and prevent obstruction. However, stent-related biofilm formation remains a significant clinical problem, contributing to infection, encrustation, patient discomfort, and stent failure. Biofilms consist of microbial communities embedded within an extracellular polymeric substance (EPS), which protects microorganisms from host defenses and antimicrobial agents.

Antibiotic therapy alone may be insufficient to eradicate established biofilms due to poor penetration into the EPS matrix. Linezolid is a potent antibiotic with activity against gram-positive organisms commonly implicated in urinary tract colonization and penetrate and effectively act against bacterial biofilms. Mucolytic agents, by disrupting the biofilm matrix, may enhance antimicrobial penetration and reduce biofilm burden.

The combination of an antibiotic with a mucolytic agent may therefore provide superior biofilm reduction compared to either approach alone or no treatment.

ELIGIBILITY:
Inclusion Criteria

* Adult patients (≥18 years).
* Undergoing lithotripsy (FURS, URS or PCNL) with DJ stent insertion.
* Stone free status.
* Planned stent indwelling time of 1 month.
* Negative preoperative urine culture.

Exclusion Criteria

* Known allergy or contraindication to linezolid or the selected mucolytic agent.
* Chronic kidney disease.
* Immunocompromised patients (e.g., chemotherapy, long-term steroid use).
* Pregnant or lactating women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Biofilm bacterial load | 1 month
  Biofilm bacterial load, defined as the quantity of bacteria within a biofilm, measured by culture of a swab taken off Double J stent after removal and expressed in numbers.

SECONDARY OUTCOMES:
Urinary tract infection rate | 1 month
  urinary tract infection, defined as presence of positive urine culture after double J stent insertion, expressed in numbers.
Double J related symptoms | 1 month
  Double J related symptoms, defined as lower urinary tract symptoms that patient expeirence after double J stent insertion, measured using the ureteral stent symptom questionnaire (USSQ), expressed in numbers.

CONTACTS AND LOCATIONS:
Locations (1):
- Menoufia Faculty of Medicine, Shebin El-Kom, Menoufia, Egypt